CLINICAL TRIAL: NCT03013621
Title: Venous Congestion and Acute Renal Failure in Cardiac Surgery Postoperative (COVD)
Brief Title: Venous Congestion and Acute Renal Failure in Cardiac Surgery Postoperative
Acronym: COVD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6296
Record Dates: First submitted 2016-08-30; First posted 2017-01-06 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2016-08

CONDITIONS: Acute Renal Failure (ARF)
Keywords: Renal Failure; Renal Insufficiency; Acute Renal Failure; Acute Renal Injury; Kidney Failure; Kidney Insufficiency; Acute Kidney Failure; Acute Kidney Injury; Ventricular dysfunction; Venous congestion; Renal function; Kidney function; Venous heart failure
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency; Ventricular Dysfunction; Hyperemia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Acute renal failure (ARF) is a frequent complication in the postoperative cardiac surgery, and is a major risk factor for mortality in this context.

The right ventricular dysfunction post cardiopulmonary bypass (CPB) is also a common complication, close to 100% if one takes into account the transient dysfunction.

A recent study showed that right ventricular dysfunction and the IRA seemed related, rather on the slope of venous congestion. We wish to study this phenomenon more specifically in particular to offer reliable diagnostic markers of venous congestion.

ELIGIBILITY:
Inclusion Criteria:

* Age: all major patient
* Gender: both
* Subject has signed an informed consent
* IRA KDIGO stage 1 or urine output <0.5 mL / kg / h for at least 6 hours / elevation creat> 26.5μmol / L
* Patient in sinus rhythm at the time of the ultrasound measurements
* No diuretic since intervention
* Absence of circulatory failure (low doses of catecholamines tolerated)
* Extubated: absence of mechanical ventilation

Exclusion Criteria:

* Chronic heart failure right
* Chronic renal failure (GFR <60)
* Usual treatment with high dose diuretics (furosemide> 40mg / day)
* Endocarditis
* Emergency surgery (aortic dissection, emergency bypass surgery) / heart surgery D / redux
* Circulatory Support
* ACFA / electro-paced rhythm
* Inability to give informed about information (subject in emergencies, understanding of the subject of difficulty, ...)
* Topic under judicial protection
* Topic guardianship or curatorship
* Pregnancy (women of childbearing age)
* Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of patients in immediate postoperative period of cardiac surgery, hospitalized in surgical intensive care department
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Quantification of sonographic markers of right ventricular | 1 hour after cardiac surgery

CONTACTS AND LOCATIONS:
Overall Officials: Paul-Michel MERTES, MD, PhD, Study Director — University Hospital, Strasbourg, France
Locations (1):
- Service Réanimation chirurgicale cardio-vasculaire - NHC, Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No